CLINICAL TRIAL: NCT06482593
Title: Periapical Healing in Response to Endodontically Treated Teeth With Different Sealing Cements: An in Vivo Study With CBCT
Brief Title: Periapical Healing in Response to Endodontically Treated Teeth With Different Sealing Cement
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institucion Universitaria Colegios de Colombia (Other)
Responsible Party: Principal Investigator, Nestor Raúl Rios Osorio, Dentistry, Specialization in Endodontics, Master in Sciences, Institucion Universitaria Colegios de Colombia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRios_Periapical-Healing_CBCT
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Apical Periodontitis
Keywords: Clinical Trial; Endodontic Sealer; Periapical healing
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Groupe 1: ZOE-based sealant (Active Comparator): ZOE-based sealant (GROSS-MAN, PROQUIDENT, COL)
  Interventions: Drug: Zinc-Oxide Eugenol Sealer
- Groupe 2: AH-Plus Epoxy Resin Sealer (Active Comparator): Epoxy resin-based sealant (AH Plus, Dentsply DeTrey, Konstanz, Germany)
  Interventions: Drug: AH-Plus Epoxy Resin Sealer
- Groupe 3: Bio-C Sealer (Experimental): Bioceramic sealer (Bio-C Sealer, ANGELUS, BRA)
  Interventions: Drug: Bio-C Sealer

INTERVENTIONS:
Drug: Zinc-Oxide Eugenol Sealer — Zinc oxide-eugenol sealers have a slow setting time, shrinkage while setting, solubility, and can discolour tooth structure. This sealer group has an advantage in terms of antibacterial activity.It will absorb if extruded into the periradicular tissues.
  Arms: Groupe 1: ZOE-based sealant
Drug: AH-Plus Epoxy Resin Sealer — Dentsply AH Plus Root Canal Sealing Material is a two-component paste/paste root canal sealer based on epoxy-amine resin. The AH Plus sealer shows extremely low shrinkage making it a suitable choice of material to seal the root canal.
  Arms: Groupe 2: AH-Plus Epoxy Resin Sealer
Drug: Bio-C Sealer — Bio-C® Sealer is a ready-to-use, bioceramic root canal sealer with biologically active ingredients to seal and heal the root canal space. Bio-C Sealer's mechanical and physical properties make it easy to manipulate and seal the canals, while its biological properties and high pH ensure safety and treatment success.
  Other Names: Bioceramic Sealer
  Arms: Groupe 3: Bio-C Sealer

SUMMARY:
The goal of this clinical trial is to conduct an in vivo study that allows to compare the periapical healing process of 3 different sealing cements through CBCT, as well as implement the evaluation of these lesions through volumetric measurements to provide high-level scientific information and thus have the possibility of being applied in the clinical dental practice, in patients attending UNICOC dental clinics between 2023 and 2024. The main question it aims to answer is:

* Do bioceramic sealer promote faster periapical healing due to their better sealing capacity and high bio-compatibility?
* Are there no differences between endodontic sealers in terms of apical healing? If there is a comparison group: Researchers will compare Bio-C Sealer (Bioceramic sealer) Zinc-oxide eugenol sealer and AH-Plus epoxy resin sealer to evaluate periapical healing after a six months follow-up of conventional endodontic therapy.

Coronal permanent restoration must be performed no later than 15 days after endodontic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60
* Patients systemically healthy (ASA I)
* Patients that require endodontic therapy for single-rooted teeth with pulp necrosis and apical periodontitis (AP).
* CBCT PAI periapical index score 3 or above, with no symptoms at the time of appointment.

Exclusion Criteria:

* Exclusion criteria included other than ASA-1 classification
* Patients with Perforated cortical plates at cbct analysis
* Premature permanent teeth
* Patients with Endodontic-periodontic lesions, dystrophic calcifications, more than 20° root curvature
* Pregnancy or lactation
* Root fracture cases
* Use of analgesics within 12-24 hours root canal therapy and patients with endodontic abscess.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric Periapical Healing | Six months follow-up
  Changes of the three-dimensional volume of the periapical lesion of endodontic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinics of the University College of Colombia, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galler KM, Weber M, Korkmaz Y, Widbiller M, Feuerer M. Inflammatory Response Mechanisms of the Dentine-Pulp Complex and the Periapical Tissues. Int J Mol Sci. 2021 Feb 2;22(3):1480. doi: 10.3390/ijms22031480. PMID 33540711
- [Background] Holland R, Gomes JE Filho, Cintra LTA, Queiroz IOA, Estrela C. Factors affecting the periapical healing process of endodontically treated teeth. J Appl Oral Sci. 2017 Sep-Oct;25(5):465-476. doi: 10.1590/1678-7757-2016-0464. PMID 29069143
- [Background] Fukada SY, Silva TA, Garlet GP, Rosa AL, da Silva JS, Cunha FQ. Factors involved in the T helper type 1 and type 2 cell commitment and osteoclast regulation in inflammatory apical diseases. Oral Microbiol Immunol. 2009 Feb;24(1):25-31. doi: 10.1111/j.1399-302X.2008.00469.x. PMID 19121066
- [Background] Neves MAS, Provenzano JC, Fonseca SCL, Rodrigues RCV, Goncalves LS, Siqueira JF Jr, Rocas IN. Disinfection and outcome of root canal treatment using single-file or multifile systems and Ca(OH)2 medication. Braz Dent J. 2020 Sep-Oct;31(5):493-498. doi: 10.1590/0103-6440202003245. PMID 33146332
- [Background] Yoneda N, Noiri Y, Matsui S, Kuremoto K, Maezono H, Ishimoto T, Nakano T, Ebisu S, Hayashi M. Development of a root canal treatment model in the rat. Sci Rep. 2017 Jun 12;7(1):3315. doi: 10.1038/s41598-017-03628-6. PMID 28607360
- [Background] Schneeweis LA, Willard D, Milla ME. Functional dissection of osteoprotegerin and its interaction with receptor activator of NF-kappaB ligand. J Biol Chem. 2005 Dec 16;280(50):41155-64. doi: 10.1074/jbc.M506366200. Epub 2005 Oct 7. PMID 16215261
- [Background] Nair PN. On the causes of persistent apical periodontitis: a review. Int Endod J. 2006 Apr;39(4):249-81. doi: 10.1111/j.1365-2591.2006.01099.x. PMID 16584489
- [Background] Vishwanath V, Rao HM. Gutta-percha in endodontics - A comprehensive review of material science. J Conserv Dent. 2019 May-Jun;22(3):216-222. doi: 10.4103/JCD.JCD_420_18. PMID 31367101
- [Background] Shanahan DJ, Duncan HF. Root canal filling using Resilon: a review. Br Dent J. 2011 Jul 22;211(2):81-8. doi: 10.1038/sj.bdj.2011.573. PMID 21779066
- [Background] Pereira TM, Piva E, Cuevas-Suarez CE, Ricci Volpato LE, Neto MDSDS, Pivatto K, Pecora JD, Borges AH. Experimental Resin-Based Monoblock Endodontic Obturation System. Biomed Res Int. 2019 Nov 7;2019:3512606. doi: 10.1155/2019/3512606. eCollection 2019. PMID 31815132
- [Background] Komabayashi T, Colmenar D, Cvach N, Bhat A, Primus C, Imai Y. Comprehensive review of current endodontic sealers. Dent Mater J. 2020 Sep 29;39(5):703-720. doi: 10.4012/dmj.2019-288. Epub 2020 Mar 24. PMID 32213767
- [Background] Eriksen HM, Orstavik D, Kerekes K. Healing of apical periodontitis after endodontic treatment using three different root canal sealers. Endod Dent Traumatol. 1988 Jun;4(3):114-7. doi: 10.1111/j.1600-9657.1988.tb00307.x. No abstract available. PMID 3248573
- [Background] Tiburcio-Machado CS, Michelon C, Zanatta FB, Gomes MS, Marin JA, Bier CA. The global prevalence of apical periodontitis: a systematic review and meta-analysis. Int Endod J. 2021 May;54(5):712-735. doi: 10.1111/iej.13467. Epub 2021 Jan 22. PMID 33378579
- [Background] Lo Giudice R, Nicita F, Puleio F, Alibrandi A, Cervino G, Lizio AS, Pantaleo G. Accuracy of Periapical Radiography and CBCT in Endodontic Evaluation. Int J Dent. 2018 Oct 16;2018:2514243. doi: 10.1155/2018/2514243. eCollection 2018. PMID 30410540
- [Background] Kruse C, Spin-Neto R, Reibel J, Wenzel A, Kirkevang LL. Diagnostic validity of periapical radiography and CBCT for assessing periapical lesions that persist after endodontic surgery. Dentomaxillofac Radiol. 2017 Oct;46(7):20170210. doi: 10.1259/dmfr.20170210. Epub 2017 Jul 14. PMID 28707526
- [Background] Jalali P, Riccobono J, Augsburger RA, Tahmasbi-Arashlow M. Radiographic patterns of periosteal bone reactions associated with endodontic lesions. Restor Dent Endod. 2023 Jun 8;48(3):e23. doi: 10.5395/rde.2023.48.e23. eCollection 2023 Aug. PMID 37675448